CLINICAL TRIAL: NCT00852956
Title: Evaluation of Safety, Drug-Drug Interactions and Pharmacokinetic Profiles of Co-Administration of Betahistine With Olanzapine in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OBEcure Ltd. (Industry)
Responsible Party: Nir Barak, OBEcure Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: OBE 209
Record Dates: First submitted 2009-02-23; First posted 2009-02-27 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: Betahistine; Olanzapine; Safety of co-administration of Betahistien and Olanzapine
MeSH Terms: interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Betahistine 48 mg TID; 08:00, 13:00 and 18:00 (144 mg/day total)and Olanzapine (10 mg/day)
  Interventions: Drug: Betahistine
- Control (Active Comparator): Matching placebo TID; 08:00, 13:00 and 18:00 and Olanzapine (10 mg/day).
  Interventions: Drug: Betahistine

INTERVENTIONS:
Drug: Betahistine — The study will be comprised of three treatment periods for a total of 4 weeks treatment duration:
  Period I 1 week (Days 1-7) administration of betahistine 48 mg three times daily (144 mg/day total) or matching placebo Period II 1 week (Days 8-14) titration of olanzapine once daily (from 2.5 mg up to 10 mg) and continuation of betahistine or matching placebo administration (three times daily as in Period I) Period III 2 weeks (Days 15-28) of co-administration of betahistine or matching placebo (three times daily; as in Periods II and III) and olanzapine once daily (7.5 or 10 mg, as tolerated)
  On Day 1, after a 7-day screening period, eligible subjects will be randomized to one of the two treatment groups in a 1:1 ratio:
  Betahistine 48 mg TID; 08:00, 13:00 and 18:00 (144 mg/day total) Matching placebo TID; 08:00, 13:00 and 18:00

SUMMARY:
This will be a phase I, randomized, two-arm, double-blind, placebo-controlled, sequential study in up to 50 healthy female subjects. The study will be comprised of three treatment periods for a total of 4 weeks treatment duration:

Period I 1 week (Days 1-7) administration of betahistine daily (three times per day; 144 mg/day total) or matching placebo.

Period II 1 week (Days 8-14) titration of olanzapine once daily (2.5 to 10 mg) and continuation of betahistine or matching placebo administration (daily; three times per day) Period III 2 weeks (Days 15-28) of continued co-administration of betahistine/matching placebo, three times per day, and olanzapine once daily (7.5 to 10 mg/day)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects 18 to 45 years of age.
2. Signed written informed consent.
3. Willing and able to comply with study procedures (including staying overnight in the research facility for required period for PK sampling).
4. Regular menstrual period.
5. All subjects should be non-lactating, have a negative urine pregnancy test result, and do not plan on become pregnant during the study, must practice or be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration.
6. Has been on a stable treatment regimen with any of the following medications for a minimum of 90 days prior to screening:

   * Hormone replacement therapy;
   * Oral contraceptives.

Exclusion Criteria:

1. Has abnormal body composition, either overweight or obesity (BMI > 27 Kg/m2) or undernourishment (BMI < 18.5 Kg/m2).
2. Has had a significant body weight loss of >4 kg in the 90 days prior to screening.
3. Pregnancy or lactation.
4. Has recently started a smoking cessation program.
5. Has known sensitivity to betahistine or olanzapine.
6. Having first degree relatives with diabetes.
7. Personal history of gestational diabetes.
8. Subjects diagnosed with polycystic ovary disease.
9. Has a clinically significant history or presence of any of the following conditions:

   * Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities
   * Diabetes mellitus (type 1 or 2)
   * Fasting blood glucose level > 100 mg/dL or HBA1c > 6.0% at screening.
   * Renal insufficiency defined as a serum creatinine >1.5 mg/dL (133 µmol/L) at screening
   * Malignant disease within 5 years of screening
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 ULN
   * Thyroid-stimulating hormone (TSH) outside of the normal range
   * Plans on having any surgery (elective or otherwise) during the course of the study
   * Has hypertension (sitting blood pressure >140/90 mmHg at screening or randomization),
   * Has hyperlipidemia (triglycerides [TG] >200 mg/dL or low-density lipoprotein cholesterol [LDL-C] >190 mg/dL),
   * History of asthma
   * History of peptic ulcers
   * History of HIV, Hepatitis B, Hepatitis C
   * Has clinical laboratory test values (chemistry, hematology, metabolic or urinalysis) judged to be clinically significant by the investigator
   * Has a physical examination or electrocardiogram (ECG) with significant abnormalities, as judged by the investigator
   * Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion could cause the subject to be noncompliant with study procedures
   * Has psychiatric or neurological disorders requiring chronic medications (e.g., antidepressants, anti-psychotic or anti anxiety agents).
   * Chronic or as needed use of antihistamines
10. Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any medications for a period of more than 3 days (with the exception of antibiotic treatment for a period of less than 7 days).
11. Has received any investigational drug within 90 days prior to screening.
12. Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or is employed by OBEcure Ltd.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary objectives are to evaluate the safety, tolerability, pharmacokinetic profiles and drug-drug interactions of betahistine and olanzapine at steady-state in healthy female subjects. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - IFE Human Pharmacology, Arad
  - IFE Human Pharmacology, Timișoara